CLINICAL TRIAL: NCT03000673
Title: A Study to Assess Safety and Tolerability of Single Oral Doses of BMS-986177 in Patients With ESRD Treated With Chronic Hemodialysis
Brief Title: A Study to Evaluate Safety of Single Doses of BMS-986177 in Patients With End Stage Renal Disease (ESRD) Treated With Hemodialysis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV010-010
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Antithrombotic
MeSH Terms: interventions — Enoxaparin; Heparin; milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Sequence 1 (Active Comparator): UFH, BMS-986177 - dose 1, BMS-986177 - dose 2, Enoxaparin
  Interventions: Drug: Enoxaparin; Drug: unfractionated heparin (UFH); Drug: BMS-986177
- Dose Sequence 2 (Active Comparator): BMS-986177 - dose 1, Enoxaparin, UFH, BMS-986177 - dose 2
  Interventions: Drug: Enoxaparin; Drug: unfractionated heparin (UFH); Drug: BMS-986177
- Dose Sequence 3 (Active Comparator): BMS-986177 - dose 2, UFH, Enoxaparin, BMS-986177 - dose 1
  Interventions: Drug: Enoxaparin; Drug: unfractionated heparin (UFH); Drug: BMS-986177
- Dose Sequence 4 (Active Comparator): Enoxaparin, BMS-986177 - dose 2, BMS-986177 - dose 1, UFH
  Interventions: Drug: Enoxaparin; Drug: unfractionated heparin (UFH); Drug: BMS-986177

INTERVENTIONS:
Drug: Enoxaparin — Specified dose of Enoxaparin on specified days
Drug: unfractionated heparin (UFH) — Specified dose of UFH on specified days
Drug: BMS-986177 — Specified dose of BMS-986177 on specified day

SUMMARY:
To investigate safety of Single Doses of BMS-986177 in Patients with End Stage Renal Disease treated with hemodialysis

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects with ESRD treated with hemodialysis 3 times a week for at least 3 months prior enrollment.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
* Women must not be breastfeeding
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) BMS-986177 plus 5 half-lives of study treatment (2 days) plus 30 days (duration of ovulatory cycle) for a total of 32 days post-treatment completion
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) BMS-986177 plus 5 half-lives of the study treatment plus 90 days (duration of sperm turnover) for a total of 92 days post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Subjects receiving dialysis through central venous catheters
* History of uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, psychiatric and/or neurological disease in the past 3 months
* Current or recent (within 3 months of study drug administration) gastrointestinal disease or surgery, which by the judgment of the Investigator, may increase a subject's risk of gastrointestinal bleeding or interfere with absorption of study drug (e.g., peptic or gastric ulcer disease, severe gastritis, history of gastrointestinal surgery).
* Any major surgery within 12 weeks of study drug administration
* History of significant head injury within the last 2 years, including subjects with base of skull fractures

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Davita Clinical Research, Lakewood, Colorado
  - Orlando Clinical Research Center, Orlando, Florida
  - Davita Clinical Research, Minneapolis, Minnesota

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 participants were randomized and treated.
Groups:
- Sequence ABCD; Sequence BDAC; Sequence CADB; Sequence DCBA: Treatments: A = UFH intravenous infusion; B = BMS-986177 100 mg; C = BMS-986177 300 mg; D = enoxaparin 40 mg by subcutaneous injection
Period: Overall Study
Arm/Group | Sequence ABCD | Sequence BDAC | Sequence CADB | Sequence DCBA
Started | 7 | 9 | 7 | 9
Completed | 6 | 9 | 7 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Seq ABCD; Seq BDAC; Seq CADB; Seq DCBA: Treatments: A=UFH intravenous infusion; B=BMS-986177 100 mg; C=BMS-986177 300 mg; D=Enoxaparin 40 mg by subcutaneous injection
- Total: Total of all reporting groups
Arm/Group | Seq ABCD | Seq BDAC | Seq CADB | Seq DCBA | Total
Number analyzed (Participants) | 7 | 9 | 7 | 9 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (7.3) | 55.6 (6.6) | 52.0 (12.4) | 51.7 (9.9) | 53.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 3 | 12
  Male | 6 | 4 | 4 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 9 | 7 | 9 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1 | 0 | 1 | 1 | 3
  Black or African American | 6 | 9 | 6 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: The Number of Adverse Events (AEs), Serious AEs (SAEs), AEs Leading to Discontinuation and Death
Description: Safety and tolerability of single oral doses of BMS-986177 in patients with end-stage renal disease (ESRD) on chronic hemodialysis (HD) treatment as measured by the number of participants with adverse events (AEs), serious AEs (SAEs), AEs leading to discontinuation and death
Time Frame: From the date of patient's written consent to participate in study until 30 days after discontinuation of dosing or patient's participation in study (up to October 2017)
Population: All treated participants
Measure: Number; unit: Participants
Groups:
- Treatment B: Treatment B = BMS-986177 100 mg oral suspension
- Treatment C: Treatment C = BMS-986177 300 mg oral suspension
- Treatment D: Treatment D = enoxaparin 40 mg by subcutaneous injection
- Treatment A: Treatments: A = UFH intravenous infusion
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
Participants
  Adverse Events | 4 | 4 | 3 | 2
  Serious Adverse Events | 0 | 0 | 0 | 0
  Adverse Events Leading to Discontinuations | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

2. Primary Outcome: The Number of Participants Marked Abnormalities in Clinical Laboratory Tests : Hematology I; Hematology II; Coagulation
Description: HEMATOLOGY I; HEMOGLOBIN HB G/DL LOW < 0.85*PRE-RX; HEMATOCRIT HCT % LOW < 0.85*PRE-RX; PLATELET COUNT PLAT X10*9 C/L LOW < 0.85*LLN IF PRE-RX IS MISSING; < 0.85*LLN IF PRE-RX >= LLN; < 0.85*PRE-RX IF PRE-RX < LLN; HIGH > 1.5*ULN; HEMATOLOGY II; LEUKOCYTES WBC X10*3 C/UL LOW < 0.9*LLN IF PRE-RX IS MISSING; < 0.9*LLN IF LLN <= PRE-RX <= ULN; < 0.85*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN; HIGH > 1.2*ULN IF PRE-RX IS MISSING; > 1.2*ULN IF LLN <= PRE-RX <= ULN; > 1.5*PRE-RX IF PRE-RX > ULN; NEUTROPHILS (ABSOLUTE) NEUTA X10*3 C/UL LOW < 1.5 IF PRE-RX IS MISSING; < 1.5 IF PRE-RX >= 1.5; < 0.85*PRE-RX IF; PRE-RX < 1.5; LYMPHOCYTES (ABSOLUTE) LYMPA X10*3 C/UL LOW < 0.75; HIGH > 7.5; MONOCYTES (ABSOLUTE) MONOA X10*3 C/UL HIGH > 2; BASOPHILS (ABSOLUTE) BASOA X10*3 C/UL HIGH > 0.4; EOSINOPHILS (ABSOLUTE) EOSA X10*3 C/UL HIGH > 0.75; COAGULATION: PROTHROMBIN TIME (PT) PT SEC HIGH > 1.5*ULN; APTT APTT SEC HIGH > 1.5*ULN; INTL NORMALIZED RATIO (INR) INR FRACTION HIGH > 1.5*ULN;
Time Frame: At screening; On Day -3 to Day -1, 3 to 6 hours post HD on Days 1, 5, 8, and 12; and at study discharge.
Population: All treated participants with evaluable test results
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
Participants
  Hematology I Hemoglobin (G/DL) Abnormal low: number analyzed (Participants) | 31 | 31 | 31 | 31
  Hematology I Hemoglobin (G/DL) Abnormal low | 3 | 3 | 2 | 1
  Hematocrit (%) Abnormal low: number analyzed (Participants) | 31 | 31 | 31 | 31
  Hematocrit (%) Abnormal low | 3 | 4 | 2 | 2
  Platelet Count (X10*9 C/L) Abnormal low: number analyzed (Participants) | 31 | 31 | 31 | 31
  Platelet Count (X10*9 C/L) Abnormal low | 1 | 1 | 2 | 1
  Leukocytes (X10*3 C/UL) Abnormal low: number analyzed (Participants) | 31 | 31 | 31 | 31
  Leukocytes (X10*3 C/UL) Abnormal low | 2 | 1 | 0 | 2
  Leukocytes (X10*3 C/UL): Abnormal high: number analyzed (Participants) | 31 | 31 | 31 | 31
  Leukocytes (X10*3 C/UL): Abnormal high | 0 | 0 | 1 | 1
  Neutrophils (Absolute) (X10*3 C/UL): number analyzed (Participants) | 31 | 31 | 31 | 31
  Neutrophils (Absolute) (X10*3 C/UL) | 0 | 0 | 2 | 1
  Lymphocytes (Absolute) (X10*3 C/UL) Abnormal low: number analyzed (Participants) | 31 | 31 | 31 | 31
  Lymphocytes (Absolute) (X10*3 C/UL) Abnormal low | 3 | 4 | 3 | 5
  Monocytes (Absolute) (X10*3 C/UL) Abnormal high: number analyzed (Participants) | 31 | 31 | 31 | 31
  Monocytes (Absolute) (X10*3 C/UL) Abnormal high | 0 | 0 | 0 | 0
  Basophils (Absolute) (X10*3 C/UL) Abnormal high: number analyzed (Participants) | 31 | 31 | 31 | 31
  Basophils (Absolute) (X10*3 C/UL) Abnormal high | 0 | 0 | 0 | 0
  Eosinophils (Absolute) (X10*3 C/UL): number analyzed (Participants) | 32 | 31 | 31 | 31
  Eosinophils (Absolute) (X10*3 C/UL) | 1 | 1 | 2 | 1
  Prothrombin time (PT) (sec): Abnormal high: number analyzed (Participants) | 31 | 31 | 31 | 32
  Prothrombin time (PT) (sec): Abnormal high | 1 | 1 | 2 | 0
  APTT (sec): Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  APTT (sec): Abnormal high | 4 | 25 | 1 | 0
  APTT (sec): Not reported: number analyzed (Participants) | 32 | 30 | 31 | 32
  APTT (sec): Not reported | 1 | 0 | 0 | 1
  INR (fraction): Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  INR (fraction): Abnormal high | 0 | 0 | 0 | 0

3. Primary Outcome: The Number of Marked Abnormalities in Clinical Laboratory Tests (Cont.) : Liver and Kidney Function
Description: LIVER & KIDNEY FUNCTION; ALKALINE PHOSPHATASE (ALP) ALP U/L HIGH > 1.25*ULN IF PRE-RX IS MISSING; > 1.25*ULN IF PRE-RX <= ULN; > 1.25*PRE-RX IF PRE-RX > ULN; ASPARTATE AMINOTRANSFERASE (AST) AST U/L HIGH > 1.25*ULN IF PRE-RX IS MISSING; > 1.25*ULN IF PRE-RX <= ULN; > 1.25*PRE-RX IF PRE-RX > ULN; ALANINE AMINOTRANSFERASE (ALT) ALT U/L HIGH > 1.25*ULN IF PRE-RX IS MISSING; > 1.25*ULN IF PRE-RX <= ULN; > 1.25*PRE-RX IF PRE-RX > ULN; BILIRUBIN, TOTAL TBILI MG/DL HIGH > 1.1*ULN IF PRE-RX IS MISSING; > 1.1*ULN IF PRE-RX <= ULN; > 1.25*PRE-RX IF PRE-RX > ULN; BILIRUBIN, DIRECT DBILI MG/DL HIGH > 1.1*ULN IF PRE-RX IS MISSING; > 1.1*ULN IF PRE-RX <= ULN; > 1.25*PRE-RX IF PRE-RX > ULN; BLOOD UREA NITROGEN BUN MG/DL HIGH > 1.1*ULN IF PRE-RX IS MISSING; > 1.1*ULN IF PRE-RX <= ULN; > 1.2*PRE-RX IF PRE-RX > ULN; CREATININE CREAT MG/DL HIGH > 1.5*ULN IF PRE-RX IS MISSING; > 1.5*ULN IF PRE-RX <= ULN; > 1.33*PRE-RX IF PRE-RX > ULN;
Time Frame: At screening; On Day -3 to Day -1, 3 to 6 hours post HD on Days 1, 5, 8, and 12; and at study discharge.
Population: All treated participants with evaluable test results
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
Participants
  ALP (U/L) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  ALP (U/L) Abnormal high | 0 | 0 | 0 | 1
  AST (U/L) Abnormal high: number analyzed (Participants) | 32 | 30 | 30 | 32
  AST (U/L) Abnormal high | 0 | 0 | 0 | 0
  AST (U/L) Not reported: number analyzed (Participants) | 32 | 31 | 30 | 32
  AST (U/L) Not reported | 0 | 0 | 1 | 0
  ALT (U/L) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  ALT (U/L) Abnormal high | 0 | 0 | 1 | 0
  Bilirubin, Total (MG/DL) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  Bilirubin, Total (MG/DL) Abnormal high | 0 | 0 | 1 | 0
  Bilirubin, Direct (MG/DL) Abnormal high: number analyzed (Participants) | 32 | 30 | 30 | 32
  Bilirubin, Direct (MG/DL) Abnormal high | 1 | 1 | 1 | 3
  Bilirubin, Direct (MG/DL), Not reported: number analyzed (Participants) | 32 | 30 | 30 | 32
  Bilirubin, Direct (MG/DL), Not reported | 1 | 0 | 1 | 0
  Blood Urea Nitrogen (MG/DL) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  Blood Urea Nitrogen (MG/DL) Abnormal high | 0 | 1 | 1 | 0
  Creatinine (MG/DL) Abnormal high: number analyzed (Participants) | 31 | 30 | 31 | 32
  Creatinine (MG/DL) Abnormal high | 0 | 0 | 0 | 0
  Creatinine (MG/DL) Not reported: number analyzed (Participants) | 31 | 30 | 31 | 32
  Creatinine (MG/DL) Not reported | 1 | 0 | 0 | 1

4. Primary Outcome: The Number of Marked Abnormalities in Clinical Laboratory Tests (Cont.): Electrolytes
Description: ELECTROLYTES: SODIUM, SERUM NA MEQ/L LOW < 0.95*LLN IF PRE-RX IS MISSING; < 0.95*LLN IF PRE-RX >= LLN; < 0.95*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN; HIGH > 1.05*ULN IF PRE-RX IS MISSING; > 1.05*ULN IF PRE-RX <= ULN; > 1.05*PRE-RX IF PRE-RX > ULN; > ULN IF PRE-RX < LLN; POTASSIUM, SERUM K MEQ/L LOW < 0.9*LLN IF PRE-RX IS MISSING; < 0.9*LLN IF PRE-RX >= LLN; < 0.9*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN; HIGH > 1.1*ULN IF PRE-RX IS MISSING; > 1.1*ULN IF PRE-RX <= ULN; > 1.1*PRE-RX IF PRE-RX > ULN; > ULN IF PRE-RX < LLN; CHLORIDE, SERUM CL MEQ/L LOW < 0.9*LLN IF PRE-RX IS MISSING; < 0.9*LLN IF PRE-RX >= LLN; < 0.9*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN; HIGH > 1.1*ULN IF PRE-RX IS MISSING; > 1.1*ULN IF PRE-RX <= ULN; > 1.1*PRE-RX IF PRE-RX > ULN; > ULN IF PRE-RX < LLN;
Time Frame: At screening; On Day -3 to Day -1, 3 to 6 hours post HD on Days 1, 5, 8, and 12; and at study discharge
Population: All treated participants with evaluable test results
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
Participants
  Sodium, Serum (MEQ/L), Abnormal low: number analyzed (Participants) | 32 | 30 | 31 | 32
  Sodium, Serum (MEQ/L), Abnormal low | 0 | 0 | 0 | 0
  Sodium, Serum (MEQ/L), Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  Sodium, Serum (MEQ/L), Abnormal high | 0 | 0 | 0 | 0
  Potassium, Serum (MEQ/L), Abnormal low: number analyzed (Participants) | 32 | 30 | 30 | 32
  Potassium, Serum (MEQ/L), Abnormal low | 0 | 0 | 0 | 0
  Potassium, Serum (MEQ/L), Abnormal high: number analyzed (Participants) | 32 | 30 | 30 | 32
  Potassium, Serum (MEQ/L), Abnormal high | 0 | 1 | 1 | 1
  Potassium, Serum (MEQ/L), Not reported: number analyzed (Participants) | 32 | 30 | 30 | 32
  Potassium, Serum (MEQ/L), Not reported | 0 | 0 | 1 | 0
  Chloride, Serum (MEQ/L) Abnormal low: number analyzed (Participants) | 32 | 30 | 31 | 32
  Chloride, Serum (MEQ/L) Abnormal low | 0 | 0 | 0 | 0
  Chloride, Serum (MEQ/L) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  Chloride, Serum (MEQ/L) Abnormal high | 0 | 0 | 0 | 0
  Chloride, Serum (MEQ/L) Not reported: number analyzed (Participants) | 32 | 30 | 31 | 32
  Chloride, Serum (MEQ/L) Not reported | 0 | 0 | 0 | 1

5. Primary Outcome: The Number of Marked Abnormalities in Clinical Laboratory Tests (Cont.): Electrolytes (Cont.)
Description: ELECTROLYTES (CONT.): CALCIUM, TOTAL CA MG/DL LOW < 0.9*LLN IF PRE-RX IS MISSING; < 0.9*LLN IF PRE-RX >= LLN; < 0.9*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN; HIGH > 1.1*ULN IF PRE-RX IS MISSING; > 1.1*ULN IF PRE-RX <= ULN; > 1.1*PRE-RX IF PRE-RX > ULN; > ULN IF PRE-RX < LLN; PHOSPHORUS, INORGANIC PHOS MG/DL LOW < 0.85*LLN IF PRE-RX IS MISSING; < 0.85*LLN IF PRE-RX >= LLN; < 0.85*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN; HIGH > 1.25*ULN IF PRE-RX IS MISSING; > 1.25*ULN IF PRE-RX <= ULN; > 1.25*PRE-RX IF PRE-RX > ULN; > ULN IF PRE-RX < LLN; MAGNESIUM, SERUM MG MEQ/L LOW < 0.9*LLN IF PRE-RX IS MISSING; < 0.9*LLN IF PRE-RX >= LLN; < 0.9*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN; HIGH > 1.1*ULN IF PRE-RX IS MISSING; > 1.1*ULN IF PRE-RX <= ULN; > 1.1*PRE-RX IF PRE-RX > ULN; > ULN IF PRE-RX < LLN
Time Frame: At screening; On Day -3 to Day -1, 3 to 6 hours post HD on Days 1, 5, 8, and 12; and at study discharge.
Population: All treated participants with evaluable test results
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
Participants
  Calcium, Total (MG/DL) Abnormal low: number analyzed (Participants) | 32 | 30 | 31 | 32
  Calcium, Total (MG/DL) Abnormal low | 0 | 0 | 0 | 1
  Calcium, Total (MG/DL) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  Calcium, Total (MG/DL) Abnormal high | 0 | 0 | 0 | 0
  Phosphorus, Inorganic (MG/DL) Abnormal low: number analyzed (Participants) | 32 | 30 | 31 | 32
  Phosphorus, Inorganic (MG/DL) Abnormal low | 0 | 1 | 1 | 2
  Phosphorus, Inorganic (MG/DL) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  Phosphorus, Inorganic (MG/DL) Abnormal high | 0 | 0 | 0 | 0
  Magnesium, Serum (MEQ/L), Abnormal low: number analyzed (Participants) | 32 | 30 | 30 | 32
  Magnesium, Serum (MEQ/L), Abnormal low | 0 | 1 | 0 | 1
  Magnesium, Serum (MEQ/L), Abnormal high: number analyzed (Participants) | 32 | 30 | 30 | 32
  Magnesium, Serum (MEQ/L), Abnormal high | 0 | 0 | 0 | 0
  Magnesium, Serum (MEQ/L), Not reported: number analyzed (Participants) | 32 | 30 | 30 | 32
  Magnesium, Serum (MEQ/L), Not reported | 0 | 0 | 1 | 0

6. Primary Outcome: The Number of Marked Abnormalities in Clinical Laboratory Tests (Cont.): Other Chemistry Testing
Description: GLUCOSE, FASTING SERUM GLUCF MG/DL LOW < 0.8*LLN IF PRE-RX IS MISSING; < 0.8*LLN IF PRE-RX >= LLN; < 0.8*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN; HIGH > 1.3*ULN IF PRE-RX IS MISSING > 1.3*ULN IF PRE-RX <= ULN; > 2*PRE-RX IF PRE-RX > ULN; > ULN IF PRE-RX < LLN; PROTEIN, TOTAL TPRO G/DL LOW < 0.9*LLN IF PRE-RX IS MISSING; < 0.9*LLN IF PRE-RX >= LLN; < 0.9*PRE-RX IF PRE-RX < LLN; < LLN IF PRE-RX > ULN HIGH > 1.1*ULN IF PRE-RX IS MISSING; > 1.1*ULN IF PRE-RX <= ULN; > 1.1*PRE-RX IF PRE-RX > ULN; > ULN IF PRE-RX < LLN; ALBUMIN ALB G/DL LOW < 0.9*LLN IF PRE-RX IS MISSING; < 0.9*LLN IF PRE-RX >= LLN; < 0.9*PRE-RX IF PRE-RX < LLN; CREATINE KINASE (CK) CK U/L HIGH > 1.5*ULN IF PRE-RX IS MISSING; > 1.5*ULN IF PRE-RX <= ULN; > 1.5*PRE-RX IF PRE-RX > ULN; URIC ACID URIC MG/DL HIGH > 1.2*ULN IF PRE-RX IS MISSING; > 1.2*ULN IF PRE-RX <= ULN; > 1.25*PRE-RX IF PRE-RX > ULN; LACTATE DEHYDR (LD) LD U/L HIGH > 1.25*ULN IF PRE-RX IS MISSING; > 1.25*ULN IF PRE-RX <= ULN; > 1.5*PRE-RX IF PRE-RX > ULN
Time Frame: At screening; On Day -3 to Day -1, 3 to 6 hours post HD on Days 1, 5, 8, and 12; and at study discharge.
Population: All treated participants with evaluable test results
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
Participants
  Glucose, Fasting serum (MG/DL) Abnormal low: number analyzed (Participants) | 32 | 30 | 31 | 32
  Glucose, Fasting serum (MG/DL) Abnormal low | 0 | 0 | 1 | 1
  Glucose, Fasting serum (MG/DL) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  Glucose, Fasting serum (MG/DL) Abnormal high | 2 | 2 | 4 | 4
  Protein, Total (G/DL) Abnormal low: number analyzed (Participants) | 32 | 30 | 31 | 32
  Protein, Total (G/DL) Abnormal low | 0 | 0 | 1 | 1
  Protein, Total (G/DL) Abnormal high: number analyzed (Participants) | 32 | 30 | 31 | 32
  Protein, Total (G/DL) Abnormal high | 0 | 0 | 0 | 0
  Albumin (G/DL) Abnormal low: number analyzed (Participants) | 32 | 30 | 31 | 32
  Albumin (G/DL) Abnormal low | 0 | 0 | 1 | 2
  Creatine Kinase (CK) (U/L) Abnormal high: number analyzed (Participants) | 32 | 30 | 30 | 32
  Creatine Kinase (CK) (U/L) Abnormal high | 0 | 0 | 0 | 0
  Creatine Kinase (CK) (U/L) Not reported: number analyzed (Participants) | 32 | 30 | 30 | 32
  Creatine Kinase (CK) (U/L) Not reported | 0 | 0 | 1 | 0
  Uric Acid (MG/DL) Abnormal High: number analyzed (Participants) | 32 | 30 | 31 | 32
  Uric Acid (MG/DL) Abnormal High | 0 | 0 | 0 | 0
  LD (U/L) Abnormal high: number analyzed (Participants) | 32 | 30 | 30 | 32
  LD (U/L) Abnormal high | 0 | 0 | 3 | 0
  LD (U/L) Not reported: number analyzed (Participants) | 32 | 30 | 30 | 32
  LD (U/L) Not reported | 0 | 0 | 1 | 0

7. Primary Outcome: The Number of Marked Abnormalities in Clinical Laboratory Tests (Cont.) : Urinalysis I, Special Studies
Description: URINALYSIS I; BLOOD, URINE UBLD N/A HIGH >= 2 IF PRE-RX IS MISSING; >= 2 IF PRE-RX < 1; >= 2 IF PRE-RX >= 1 SPECIAL STUDIES; OCCULT BLOOD SCREEN, FECES OCBLD N/A HIGH NEGATIVE PRE-RX CHANGING TO POSITIVE
Time Frame: At screening; On Day -3 to Day -1, 3 to 6 hours post HD on Days 1, 5, 8, and 12; and at study discharge.
Population: All treated participants with evaluable test results
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
Participants
  Blood, Urine (N/A) Abnormal high: number analyzed (Participants) | 7 | 8 | 6 | 6
  Blood, Urine (N/A) Abnormal high | 1 | 1 | 0 | 0
  Occult Blood Screen, Feces (N/A) Abnormal high: number analyzed (Participants) | 21 | 18 | 15 | 19
  Occult Blood Screen, Feces (N/A) Abnormal high | 0 | 0 | 0 | 0

8. Primary Outcome: The Change From Baseline in Electrocardiogram (ECG) Parameters: Mean Heart Rate
Description: Baseline = Last non-missing result with a collection date-time less than the date-time of the first active dose of study medication.
Time Frame: Days -3 to -1, Days 1, 5, 8, and 12.
Population: All treated participants
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
Beats/min
  Day 1: number analyzed (Participants) | 9 | 7 | 9 | 7
  Day 1 | 1.8 (8.6) | 1.4 (5.1) | 0.4 (8.1) | -0.1 (5.4)
  Day 5: number analyzed (Participants) | 7 | 9 | 9 | 7
  Day 5 | -2.1 (6.9) | 2.0 (10.8) | 2.0 (8.1) | 1.6 (5.9)
  Day 8: number analyzed (Participants) | 9 | 6 | 7 | 9
  Day 8 | 0.0 (6.9) | -2.8 (6.1) | 2.3 (4.7) | 4.0 (9.8)
  Day 12: number analyzed (Participants) | 7 | 9 | 6 | 9
  Day 12 | 0.4 (6.0) | 3.9 (9.5) | 0.8 (2.9) | 1.4 (9.5)

9. Primary Outcome: The Change From Baseline in Electrocardiogram (ECG) Parameters: PR Interval, Aggregate
Description: as for outcome 8
Time Frame: Days -3 to -1, Days 1, 5, 8, and 12.
Population: All treated participants
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
msec
  Day 1: number analyzed (Participants) | 9 | 7 | 9 | 7
  Day 1 | -1.3 (9.9) | -25.0 (67.8) | -6.9 (12.6) | 13.6 (26.3)
  Day 5: number analyzed (Participants) | 7 | 9 | 9 | 9
  Day 5 | 12.6 (21.2) | -5.8 (8.9) | -5.1 (11.8) | -25.4 (66.5)
  Day 8: number analyzed (Participants) | 9 | 6 | 7 | 9
  Day 8 | -1.2 (19.3) | 12.7 (25.5) | -22.6 (70.3) | -3.4 (27.2)
  Day 12: number analyzed (Participants) | 7 | 9 | 6 | 9
  Day 12 | -27.7 (67.9) | -5.6 (8.7) | 8.8 (12.4) | -2.6 (8.7)

10. Primary Outcome: The Change From Baseline in Electrocardiogram (ECG) Parameters: QRS Duration, Aggregate
Description: as for outcome 8
Time Frame: Days -3 to -1, Days 1, 5, 8, and 12.
Population: All treated participants
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
msec
  Day 1: number analyzed (Participants) | 9 | 7 | 9 | 7
  Day 1 | -1.1 (6.7) | 5.7 (6.2) | -0.2 (3.3) | -3.1 (11.0)
  Day 5: number analyzed (Participants) | 7 | 9 | 9 | 7
  Day 5 | -0.3 (14.8) | -0.2 (4.6) | -0.2 (4.6) | 0.6 (4.8)
  Day 8: number analyzed (Participants) | 9 | 6 | 7 | 9
  Day 8 | -0.2 (4.2) | -1.8 (8.8) | -0.7 (6.0) | 0.3 (8.6)
  Day 12: number analyzed (Participants) | 7 | 9 | 6 | 9
  Day 12 | 0.9 (6.3) | -0.1 (9.3) | -0.7 (9.7) | 2.0 (7.0)

11. Primary Outcome: The Change From Baseline in Electrocardiogram (ECG) Parameters: QT Interval, Aggregate
Description: as for outcome 8
Time Frame: Days -3 to -1, Days 1, 5, 8, and 12.
Population: All treated participants
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
msec
  Day 1: number analyzed (Participants) | 9 | 7 | 9 | 7
  Day 1 | -3.7 (22.2) | -1.6 (20.8) | -3.1 (24.0) | 3.9 (23.2)
  Day 5: number analyzed (Participants) | 7 | 9 | 9 | 7
  Day 5 | 8.4 (19.3) | -7.4 (20.1) | -2.8 (22.0) | 5.6 (15.9)
  Day 8: number analyzed (Participants) | 9 | 6 | 7 | 9
  Day 8 | -1.8 (21.3) | 12.0 (11.9) | -3.6 (24.0) | -7.4 (26.8)
  Day 12: number analyzed (Participants) | 7 | 9 | 6 | 9
  Day 12 | 0.7 (20.1) | -14.9 (28.2) | -0.7 (10.8) | -2.2 (20.4)

12. Primary Outcome: The Change From Baseline in Electrocardiogram (ECG) Parameters: QTcF Interval, Aggregate
Description: QTcF = QT corrected for heart rate using the Fridericia formula Baseline = Last non-missing result with a collection date-time less than the date-time of the first active dose of study medication.
Time Frame: Days -3 to -1, Days 1, 5, 8, and 12
Population: All treated participants
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
msec
  Day 1: number analyzed (Participants) | 9 | 7 | 9 | 7
  Day 1 | -3.2 (15.3) | 1.7 (13.5) | -1.0 (16.5) | 5.7 (15.7)
  Day 5: number analyzed (Participants) | 7 | 9 | 9 | 7
  Day 5 | 5.1 (7.6) | -4.9 (11.8) | -0.6 (13.1) | 9.9 (14.7)
  Day 8: number analyzed (Participants) | 9 | 6 | 7 | 9
  Day 8 | -1.3 (17.1) | 6.2 (6.7) | 0.3 (19.7) | -2.1 (18.5)
  Day 12: number analyzed (Participants) | 7 | 9 | 6 | 9
  Day 12 | 2.1 (15.0) | -9.9 (22.8) | 0.8 (7.1) | 1.0 (10.5)

13. Primary Outcome: The Change From Baseline in Vital Signs: Diastolic Blood Pressure
Time Frame: Days -3 to -1, 1, 5, 8, 12 and at study discharge on day 13 to day 15
Population: All treated participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
mmHg
  3 hours post Hemodialysis: number analyzed (Participants) | 32 | 31 | 30 | 32
  3 hours post Hemodialysis | -3.7 (10.5) | 0.2 (10.9) | 0.1 (9.0) | 0.5 (9.3)
  24 hours post dose: number analyzed (Participants) | 30 | 30 | 31 | 32
  24 hours post dose | -2.8 (9.9) | -2.2 (8.7) | NA (NA) — No dose of BMS-986177, as Treatment D was Enoxaparin 40 mg by subcutaneous injection | NA (NA) — No dose of BMS-986177, as Treatment A was UFH intravenous infusion

14. Primary Outcome: The Change From Baseline in Vital Signs: Systolic Blood Pressure (mm Hg)
Time Frame: Days -3 to -1, 1, 5, 8, 12 and at study discharge on day 13 to day 15
Population: All treated participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
mmHg
  3 hours post hemodialysis: number analyzed (Participants) | 32 | 31 | 30 | 32
  3 hours post hemodialysis | -6.6 (28.2) | 1.1 (24.9) | -0.2 (17.0) | -5.8 (18.0)
  24 hours post dose: number analyzed (Participants) | 30 | 30 | 31 | 32
  24 hours post dose | -8.4 (23.7) | -9.2 (17.6) | NA (NA) — No dose of BMS-986177 as Treatment D was Enoxaparin 40 mg by subcutaneous injection | NA (NA) — No dose of BMS-986177, as Treatment A was UFH intravenous infusion

15. Secondary Outcome: Pharmacokinetic Parameters of BMS-986177: Cmax
Description: Cmax: Maximum observed plasma concentration
Time Frame: Either Day 1, 5, 8, or 12 depending on the randomization sequence
Population: All treated and evaluable participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 32 | 31
ng/mL | 1120 (391.8) | 3342 (922.2)

16. Primary Outcome: The Change From Baseline in Vital Signs: Heart Rate (Beats/Min)
Time Frame: Days -3 to -1, 1, 5, 8, 12 and at study discharge on day 13 to day 15
Population: All treated participants
Measure: Mean (Standard Deviation); unit: beats/min
Groups:
- Treatment A: Treatment A = UFH intravenous infusion
Arm/Group | Treatment B | Treatment C | Treatment D | Treatment A
Number analyzed (Participants) | 32 | 31 | 31 | 32
beats/min
  3 hours post hemodialysis: number analyzed (Participants) | 32 | 30 | 30 | 32
  3 hours post hemodialysis | 4.9 (9.4) | 4.0 (7.4) | 4.5 (6.5) | 3.3 (8.9)
  24 hours post dose: number analyzed (Participants) | 30 | 30 | 31 | 32
  24 hours post dose | 4.2 (5.6) | 1.1 (7.0) | NA (NA) — No dose of BMS-986177 as Treatment D was Enoxaparin 40 mg by subcutaneous injection | NA (NA) — No dose of BMS-986177, as Treatment A was UFH intravenous infusion

17. Secondary Outcome: Pharmacokinetic Parameters of BMS-986177: Tmax
Description: Time of maximum observed plasma concentration
Time Frame: Either Day 1, 5, 8, or 12 depending on the randomization sequence
Population: All treated and evaluable participants
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 32 | 31
h | 4.531 (0.933) | 4.855 (1.042)

18. Secondary Outcome: Pharmacokinetic Parameters of BMS-986177: Area Under the Concentration Curve AUC (0-T), AUC (0-24)
Description: AUC(0-T) Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration AUC(0-24) Area under the plasma concentration-time curve from time zero to 24 hours
Time Frame: Either Day 1, 5, 8, or 12 depending on the randomization sequence
Population: All treated and evaluable participants
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 32 | 31
ng.h/mL
  AUC (0-T) | 10406.6 (4551.7) | 36112.9 (19802.5)
  AUC (0-24): number analyzed (Participants) | 30 | 31
  AUC (0-24) | 10533.4 (4492.8) | 34028.0 (12191.9)

19. Secondary Outcome: Pharmacokinetic Parameters of BMS-986177: fu
Description: Fraction of unbound drug
Time Frame: Either Day 1, 5, 8, or 12 depending on the randomization sequence
Population: All treated and evaluable participants
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 32 | 31
Percentage | 7.644 (1.257) | 7.868 (1.481)

20. Secondary Outcome: Pharmacokinetic Parameters of BMS-986177: Cmaxfu
Description: Maximum observed plasma concentration of free drug
Time Frame: Either Day 1, 5, 8, or 12 depending on the randomization sequence
Population: All treated and evaluable participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 32 | 31
ng/mL | 84.32 (30.14) | 257.9 (70.40)

21. Secondary Outcome: Pharmacokinetic Parameters of BMS-986177: Area Under the Concentration Curve AUC (0-T)fu
Description: AUC(0-T)fu Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration of free drug
Time Frame: Either Day 1, 5, 8, or 12 depending on the randomization sequence
Population: All treated and evaluable participants
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 32 | 31
ng.h/mL | 783.5 (342.1) | 2782.2 (1537.7)

22. Secondary Outcome: Pharmacokinetic Parameters of BMS-986177: Area Under the Concentration Curve AUC (3-7)
Description: AUC (3-7) : Area under the plasma concentration-time curve from 3 to 7 hours (ie, during dialysis.
  Determined from blood samples entering and exiting the dialyzer)
Time Frame: Either Day 1, 5, 8, or 12 depending on the randomization sequence
Population: All treated and evaluable participants
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Treatment B | Treatment C
Number analyzed (Participants) | 32 | 31
ng.h/mL | 2847.4 (1039.1) | 8558.1 (2509.1)

ADVERSE EVENTS:
Time Frame: From the date of the patient's written consent to participate in the study until 30 days after discontinuation of dosing
Description: The collection of nonserious AE information began 3 hours prior to dialysis start on Day 1, and continued until the follow-up contact
Groups:
- Treatment A: Treatment A = UFH intravenous infusion;
- Treatment B: Treatment B = BMS-986177 100 mg
- Treatment C: Treatment C = BMS-986177 300 mg
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03000673/Prot_002.pdf
  • Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT03000673/SAP_003.pdf